CLINICAL TRIAL: NCT01629875
Title: Efficacy and Safety of DWP450 Compared With Botox in Patients With Moderate to Severe Glabellar Line: Active Controlled, Double-blind, Randomized, Multi-center, Phase I/III Clinical Trial
Brief Title: Efficacy and Safety of DWP450 Compared With Botox in Moderate to Severe Glabellar Line
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP450001
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Moderate to Severe Glabellar Line
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- DWP450 (Experimental)
  Interventions: Drug: Generic equivalent of Clostridium Botulinum A Toxin
- Botox (Active Comparator)
  Interventions: Drug: Botox (Clostridium Botulinum A Toxin)

INTERVENTIONS:
Drug: Generic equivalent of Clostridium Botulinum A Toxin
  Arms: DWP450
Drug: Botox (Clostridium Botulinum A Toxin)
  Arms: Botox

SUMMARY:
The purpose of this study was to observe Efficacy and safety of DWP450 compared with Botox in moderate to severe glabellar line patients.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
At 4 weeks, Glabellar line improvement rate at maximum frown confirmed with investigator's live severity assessment | At 4 weeks
  At 4 weeks, Glabellar line improvement rate at maximum frown confirmed with investigator's live severity assessment

SECONDARY OUTCOMES:
At 8, 12, 16 weeks, Glabellar line improvement rate at maximum frown confirmed with investigator's live severity assessment | At 8, 12, 16 weeks
  At 8, 12, 16 weeks, Glabellar line improvement rate at maximum frown confirmed with investigator's live severity assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea